CLINICAL TRIAL: NCT02601885
Title: An Escalating Multiple Dose Study of ABT-555 in Subjects With Relapsing Forms of Multiple Sclerosis
Brief Title: A Multiple Dose Study of ABT-555 in Subjects With Relapsing Forms of Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M14-173
Record Dates: First submitted 2015-11-05; First posted 2015-11-11 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing-remitting; Secondary progressive; Relapsing forms
MeSH Terms: conditions — Multiple Sclerosis | interventions — elezanumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 2 (Experimental): Participants will receive multiple doses of ABT-555 or placebo
  Interventions: Drug: ABT-555; Other: Placebo
- Group 3 (Experimental): Participants will receive multiple doses of ABT-555 or placebo
  Interventions: Drug: ABT-555; Other: Placebo
- Group 1 (Experimental): Participants will receive multiple doses of ABT-555 or placebo
  Interventions: Drug: ABT-555; Other: Placebo

INTERVENTIONS:
Drug: ABT-555 — Intravenous Infusion
  Other Names: Elezanumab
Other: Placebo — Intravenous Infusion

SUMMARY:
This study seeks to evaluate the safety, tolerability, pharmacokinetics (PK) and immunogenicity of ABT-555 in participants with relapsing forms of multiple sclerosis (RFMS).

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving one of the following MS medications for at least 3 months: beta-interferon (any formulation including the pegylated form), glatiramer acetate (Copaxone®, others), teriflunomide (Aubagio®), fingolimod (Gilenya®), or dimethyl fumarate (Tecfidera®); OR
* Has not been treated with an MS immunotherapy for the past 6 months (12 months if they previously received cyclophosphamide or alemtuzumab); OR
* Treatment naïve with established MS diagnosis per criteria by a neurologist.
* Diagnosis of relapsing-remitting MS (RRMS) or secondary progressive MS (SPMS) according to revised McDonald criteria
* Baseline Expanded Disability Status Scale (EDSS) between 0 and 6.0, inclusive.
* Brain MRI scan at Screening that did not show evidence of overt vascular lesions, masses, mass effect or other abnormalities other than those compatible with MS, which would preclude the participant from undergoing a lumbar puncture/spinal tap for CSF collection

Exclusion Criteria:

* Diagnosis of primary progressive MS.
* Anticipated maintenance immunomodulator change, either agent or dose
* An MS relapse that occurred within the 30 days prior to randomization AND/OR the participant has not stabilized from a previous relapse prior to randomization
* Participants for whom MRI is contraindicated
* Participants who have claustrophobia that cannot be medically managed or are unable to lie still for 1 hour or more for the imaging procedures
* Findings on brain MRI scan indicating any clinically significant brain abnormality other than MS
* Contraindication for lumbar puncture

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants reporting adverse events | Throughout study from Day 1 to Day 176
Concentration of anti-drug antibody (ADA) titers of ABT-555 | Day 1 to Day 176
Time to Maximum observed plasma concentration (Tmax) of ABT-555 | Day 1 to Day 176
Maximum observed plasma concentration (Cmax) of ABT-555 | Day 1 to Day 176
Area under the concentration curve (AUC) of ABT-555 | Day 1 to Day 176

SECONDARY OUTCOMES:
Percentage of participants who experience relapse and disability progression | Throughout the study to Day 176
Lesion volume of new, newly enlarging T2 hyperintense lesions | Throughout study from Day 0 to Day 113
Number of new, newly-enlarging T2 hyperintense lesions | Throughout study from Day 0 to Day 113
Total number of new Gadolinium-enhancing T1 lesions | Throughout study from Day 0 to Day 113

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (8):
- United States (8):
  - Compass Research LLC, Orlando, Florida
  - Rowe Neurology Institute, Lenexa, Kansas
  - Parexel International, Baltimore, Maryland
  - MIND, Farmington Hills, Michigan
  - Duke Univ Med Ctr, Durham, North Carolina
  - Tri-State Mountain Neurology, Johnson City, Tennessee
  - Clinical Trial Network, Houston, Texas
  - Integrated Neurology Services, Alexandria, Virginia

IPD SHARING:
Plan to Share IPD: Undecided